CLINICAL TRIAL: NCT04935138
Title: Cell-free DNA Analysis of Chromosome Anomalies in Early Pregnancy Loss
Status: Terminated | Type: Observational
Why Stopped: Low participation
Sponsor: Quest Diagnostics-Nichols Insitute (Industry)
Collaborators: Illumina, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CD20-011
Record Dates: First submitted 2021-06-15; First posted 2021-06-22 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Early Pregnancy Loss
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: cfDNA analysis — sequencing data from cfDNA analysis

SUMMARY:
The study assesses the accuracy of cell-free DNA (cfDNA) analysis in detecting whole chromosomal aneuploidies from maternal plasma of patients with early, missed miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* 5-20 weeks of gestation by ultrasound
* Miscarriage diagnosed by ultrasound
* Pregnancy tissue still present in utero, including an empty sac, and not completely expelled

Exclusion Criteria:

* Maternal age < 18 years
* No visible pregnancy tissue on ultrasound
* Multiple fetal gestation (> than singleton)
* Pregnancy was conceived using in vitro fertilization (IVF) with preimplantation genetic testing for aneuploidy (PGT-A) performed on the transferred embryo
* No microarray testing is planned on the product of conception
* Previous normal non-invasive prenatal testing (NIPT) or diagnostic testing (chorionic villous sampling or amniocentesis) in the current pregnancy
* Patient unable to provide consent

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Previously pregnant women that have recently miscarried.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
microarray analysis of products of conception (POC) | 7 days
  chromosome anomalies

CONTACTS AND LOCATIONS:
Overall Officials: Pranoot X Tanpaiboon, MD, Principal Investigator — Quest Diagnostics-Nichols Insitute; Karen E Racicot, PhD, Principal Investigator — Quest Diagnostics-Nichols Insitute
Locations (1):
- Quest Diagnostics, San Juan Capistrano, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Practice Committee of the American Society for Reproductive Medicine. Evaluation and treatment of recurrent pregnancy loss: a committee opinion. Fertil Steril. 2012 Nov;98(5):1103-11. doi: 10.1016/j.fertnstert.2012.06.048. Epub 2012 Jul 24. PMID 22835448
- [Background] Barisic I, Zergollern L, Muzinic D, Hitrec V. Risk estimates for balanced reciprocal translocation carriers--prenatal diagnosis experience. Clin Genet. 1996 Mar;49(3):145-51. doi: 10.1111/j.1399-0004.1996.tb03274.x. PMID 8737980
- [Background] ESHRE. European Society of Human Reproduction and Embryology guideline: recurrent pregnancy loss. Human Reproduction Open 2018: 1-12.
- [Derived] Kutteh WH, Miller CE, Park JK, Corey V, Chavez M, Racicot K, Alagia DP 3rd, Jinnett KN, Curnow K, Dalton K, Bhatt S, Keefe DL. Cell-Free DNA Analysis of Fetal Aneuploidies in Early Pregnancy Loss. J Clin Med. 2024 Jul 23;13(15):4283. doi: 10.3390/jcm13154283. PMID 39124551